CLINICAL TRIAL: NCT00484471
Title: A Double Blind, Randomized, Placebo Controlled Trial of Aripiprazole Plus Valproate in the Short-Term and Long-Term Treatment of Bipolar Disorder
Brief Title: ABLE: Abilify in Bipolar Disorder for Long-term Effectiveness
Acronym: ABLE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea Otsuka International Asia Arab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 031-OTB-0701
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: aripiprazole; Drug: valproate
- 2 (Placebo Comparator)
  Interventions: Drug: valproate; Drug: placebo

INTERVENTIONS:
Drug: aripiprazole — 15-30 mg/day aripiprazole, 22 weeks
  Other Names: Abilify
  Arms: 1
Drug: valproate — sufficient dose as determined by investigator to maintain the therapeutic level.
Drug: placebo — placebo to aripiprazole, 22 weeks
  Arms: 2

SUMMARY:
To compare combination treatment of aripiprazole plus valproate versus valproate alone in the prevention of relapse in bipolar I disorder patients with symptomatic remission after 5-6 weeks open-label acute treatment with aripiprazole plus valproate for manic or mixed episode, with or without psychotic features.

DETAILED DESCRIPTION:
Further study details as provided by Korea OIAA

ELIGIBILITY:
Inclusion Criteria:

1. Subjects able to give informed consent, and/or consent obtained from a legally acceptable representative (as required by IRB/IEC) prior to the initiation of any protocol required procedures;
2. Subjects with Bipolar I Disorder, manic or mixed episode, with or without psychotic features, as defined by DSM-IV-TR and confirmed by the M.I.N.I.;
3. Subjects who are able to understand the nature of the study and follow protocol requirements including the prescribed dosage regimens, capsule/tablet ingestion, discontinuation of prohibited concomitant medications, and who can be reliably rated on assessment scales;
4. Subjects willing to discontinue all medication starting from the signing of the informed consent and during the study phases (allowed exceptions noted in Section 6.4.2);
5. Men or women aged ≥ 18 and ≤ 65 years;
6. Subjects with YMRS total score ≥ 20 (to be assessed prior entry into open-label acute treatment phase);
7. YMRS total score ≤ 12 for 2 consecutive visits (to be assessed at Week 5 and/or Week6 prior entry into double-blind treatment phase).

Exclusion Criteria:

1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to four weeks after completion of the study. Acceptable methods include oral, injectable or implanted contraceptives, intrauterine devices or barrier methods such as condoms, diaphragm, and spermicides;
2. Women who are pregnant or breast-feeding;
3. Subjects presenting clinically with a current DSM-IV-TR diagnosis of delirium, dementia, amnestic or other cognitive disorders, or a psychotic disorder (e.g., schizophrenia or schizoaffective disorder). Also, subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder;
4. Subjects with a current Axis I (DSM-IV-TR) diagnosis of Bipolar II Disorder, rapid cyclers (experiencing four or more manic or depressive episodes per year), Bipolar Disorder NOS, or any other primary psychiatric disorder other than Bipolar I Disorder;
5. Subjects with documented evidence of first manic episode;
6. Subjects considered treatment refractory for manic symptoms; (Note: if a subject has failed ≥ 2 antimanic treatments, e.g., antipsychotic, lithium, valproate or carbamazepine at therapeutic dose and duration, exclusive of the current episode, obtain permission from the Otsuka medical monitor to include the subject)
7. Subjects previously nonresponsive to aripiprazole for manic symptoms;
8. Subjects with a significant risk of committing suicide based on history, mental status exam, or investigator's judgment;
9. Subjects who have met DSM-IV-TR criteria for substance abuse within the past three months, or substance dependence* within the past 6 months, including benzodiazepines; (* exceptional for subjects with substance dependence on nicotine or caffeine);
10. Subjects with thyroid pathology (e.g., hypothyroidism or hyperthyroidism) unless condition has been stabilized with medications for at least the past three months; (Note: Subjects with an abnormal thyroid function test may be retested prior to the start of study medication. Subjects with an abnormal thyroid function test at screening will not be eligible for the study, unless permission is obtained from Otsuka);
11. Subjects who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event or interfere with assessments of safety or efficacy during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine (e.g., Addison's Disease), immune, neurologic, or hematologic disease as determined by the clinical judgment of the investigator;
12. Subjects with a significant history of seizure disorder (e.g., epilepsy);
13. The following laboratory tests results, vital signs, and ECG findings are exclusionary:

    * Platelets ≤ 75000/mm3
    * Hemoglobin ≤ 9g/dL
    * Neutrophils, absolute ≤ 1000/ mm3
    * SGOT (AST) > 3x Upper Limit of Normal
    * SGPT (ALT) > 3x Upper Limit of Normal
    * Creatinine ≥ 2 mg/dL
    * QTc > 475 msec
14. Subjects with a recent antipsychotic use who have a CPK ≥ 550 IU (Otsuka should be contacted to discuss any elevated CPK levels);
15. Subjects who are known to be allergic, intolerant, or unresponsive to valproate or to aripiprazole;
16. Subjects with a history of neuroleptic malignant syndrome from antipsychotic agents;
17. Subjects likely to require prohibited concomitant therapy during the study as indicated in Section 6.4 of the protocol;
18. Recent treatment of their most recent manic or mixed acute episode with a long acting antipsychotic in which the last dose was less than one full cycle plus one week prior to entering Phase 2 (haloperidol decanoate treatment within the past five weeks, fluphenazine decanoate treatment within the past three weeks or Risperdal ConstaTM treatment within the past three weeks);
19. Subjects likely to require the initiation of intensive individual psychotherapy during the course of the study (Note: Group and supportive therapy is allowed, if part of the subject's ongoing treatment. Individual psychotherapy is allowed if the subject has consistently received psychotherapy for at least 3 months prior to the study and will continue during the study);
20. ECT treatment within the current episode or within two months prior to the study;
21. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-10; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Time to relapse in double-blind treatment phase | throughout the study

SECONDARY OUTCOMES:
Mean change from baseline to all time point in YMRS total score; | throughout the study
Mean change from baseline to all time points in MADRS total score | throughout the study
Response rate (≥ 50% improvement in YMRS total score) at all time points | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Nan-Ying Chiu, MD, Study Chair — Changhua Christian Hospital, Taiwan; Hun-Yu Chang, MD, Principal Investigator — Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan; Yen-Kung Yang, MD, Principal Investigator — National Cheng-Kung University Hospital; Wen-Chen Ouyang, MD, Principal Investigator — Jia-Nan Mental Hospital; Wei-Wen Lin, MD, Principal Investigator — Tri-Service General Hospital; Tso-Ren Wang, MD, Principal Investigator — Tsao-Tun Psychistric Center; Efren Reyes, MD, Principal Investigator — National Center for Mental Health (NCMH); Rosanna de Guzman, MD, Principal Investigator — Philippine General Hospital (PGH); Gabino Ranoa, MD, Principal Investigator — University of Sto. Tomas Hospital (USTH); Amadeo Alinea, Principal Investigator — Veterans Medical Memorial Center (VMMC); .Vasu Chantarasak, MD, Principal Investigator — Somdej Chaophraya Hospital; Suttiporn Janenawasin, MD, Principal Investigator — Siriraj Hospital; F K Tsang, MD, Principal Investigator — Castle Peak Hospital
Locations (13):
- Castle Peak Hospital, Tuenmen, Hong Kong
- Philippines (4):
  - National Center for Mental Health, Mandaluyong
  - Philippine General Hospital, Manila
  - University of Sto. Tomas Hospital, Manila
  - Veterans Medical Memorial Center, Quezon
- Taiwan (6):
  - Changhua Chrisitian Hospital, Changhua
  - Tsao-Tun Psychiatric Center, Nantou City
  - Jia-Nan Mental Hospital, Tainan
  - National Cheng-Kung University Hospital, Tainan
  - Tri-Service General Hospital, Taipei
  - Taoyuan Mental Hospital, Taoyuan District
- Thailand (2):
  - Siriraj Hospital, Bangkok
  - Somdej Chaophraya Hospital, Bangkok